CLINICAL TRIAL: NCT03669354
Title: Spinal Manipulation Services vs. Prescription Drug Therapy for Long-term Care of Aged Medicare Beneficiaries With Chronic Low Back Pain
Brief Title: Spinal Manipulation Services vs. Prescription Drug Therapy for Long-term Care
Status: Completed | Type: Observational
Sponsor: Southern California University of Health Sciences (Other)
Collaborators: Dartmouth College (Other)
Responsible Party: Principal Investigator, Anupama KizhakkeVeettil, Professor, Southern California University of Health Sciences
Other Study IDs: 1R15AT010035-01 (NIH)
Record Dates: First submitted 2018-05-30; First posted 2018-09-13 (Actual); Results first posted 2021-09-23 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Low Back Pain
Keywords: Prescription Drugs; Spinal Manipulation
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cohort SMT: Initiation in 2013 of long-term management with SMT, and no OAT for 12 months after initiating SMT
- Cohort OAT: Initiation in 2013 of long-term management with OAT, and no SMT for 12 months after initiating OAT
- Cohort SMTX: Any occurrence of SMT for cLBP in 2013, followed by initiation in 2013 of long-term management with OAT
- Cohort OATX: Any occurrence of OAT for cLBP in 2013, followed by initiation in 2013 of long-term management with SMT

SUMMARY:
Our overall objective is to assess the value of Spinal Manipulation Services as compared to Prescription Drug Therapy for long-term management of chronic Law back Pain (LBP). Our central hypothesis is that among aged Medicare beneficiaries with chronic LBP, utilization of SMS offers superior value (to both patient and payer) for long-term care as compared to PDT.

DETAILED DESCRIPTION:
Research Design

This description applies to project specific aim 2.

Overview of Design and Methods: FFS Medicare beneficiaries will be surveyed and compared by cohort for differences in response. Subjects will be randomly sampled from each of the four cohorts (A, B, A2B & B2A) identified in SA1.

Survey Instrument and Question Formulation: A validated survey instrument will be used to collect subjective patient data. The survey will include questionnaires intended to evaluate 1) self-reported QOL, 2) satisfaction with care, and 3) beliefs regarding back pain and its treatment. For assessment of self-reported QOL a version of the SF12 (Ware '96) will be used and modified to account for time lapse between treatment for LBP and administration of the survey, and to elicit treatment-specific responses The SF -12 has been previously validated for measuring QOL among elderly patients, (Jakobsson '07) and patients using prescription drugs. (Naveiro-Rilo '14) For assessment of satisfaction with care a 0-10 numeric scale will be used. For assessment of beliefs a modified version of the validated LBP Treatment Beliefs Questionnaire will be used. (Dima '15). A pre- test of all the survey instruments will be conducted by distributing a prototype to a sample of 100 Medicare beneficiaries seen for LBP at the SCU Health Center in Whittier, CA. Responses to the survey pre-test will inform any need to edit the questionnaire for comprehensibility and ease of use, thus helping to ensure instrument face validity. For ease of comprehension by older subjects, the survey questions will be printed in large font and will be carefully worded to be brief, unambiguous, and free of bias.

Survey Methods: ResDAC will initiate contact with random samples of beneficiaries who meet criteria for inclusion in the cohorts identified in SA1. The Beneficiary Contact Service has reviewed the survey plan with the PIs and provided an official cost estimate for this service, which is routinely provided by the BCS with strict attention to patient protection. Initial contact will be in the form of a Beneficiary Notification Letter, signed by the CMS Privacy Officer. The letter will alert beneficiaries to the opportunity to voluntarily participate in a healthcare survey. Recipients will be informed that they may decline participation via enclosed reply forms, and will be given phone numbers to call CMS personnel for additional information. After three weeks, the Beneficiary Contact Service will supply the investigators with contact information for eligible beneficiaries (those who did not decline to participate). The survey will be commenced by mailing the printed survey, cover letter with informed consent form based on NCCIH guidelines, and a postage-paid return envelope with detailed information about the survey. Participants can contact study personnel if they have any questions. Follow up by phone after every two weeks or as needed will be used to increase the rate of response.

Outcomes Measurement and Statistical Analysis: Testing will be done for between-cohort differences in self-reported QOL, satisfaction with care, and beliefs about treatments for LBP. Survey responses between the four groups will be compared using Pearson chi-square tests and ANOVA. Demographic characteristics [e.g. sex as a biological variable, and age - because age-related cognitive decline can affect survey responses (Wolinsky '15)] will be controlled using linear regression for continuous survey items, proportional odds logistic regression for ordinal items and multinomial regression for categorical items. In the multivariable regression models equivalence between the four groups will be evaluated using likelihood ratio or Wald tests. Given the multiplicity of testing (e.g. multiple groups for multiple items), type I error inflation will be considered through used of Bonferonni corrections or approaches for false discovery rates. Parametric tests of numeric data can be used to yield unbiased answers when analyzing Likert scale responses. (Norman '10)

ELIGIBILITY:
Inclusion Criteria:

- Subjects will include Medicare Fee for Service beneficiaries (male or female), aged 65-84 years, residing in the US, and enrolled under Medicare Parts A, B, and D who have experienced an episode of chronic low back pain (defined as lasting three months or longer).

Exclusion Criteria:

* Subjects with diagnosis of cancer will be excluded from the study population to avoid confounding of the reason for use of prescription opioids. Subjects over the age of 85 will also be excluded.

Ages: 64 Years to 84 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The target demographic is 65-84 year old Medicare beneficiaries who were treated for at least one episode of low back pain and were enrolled in Medicare Parts A, B, and D.
Sampling Method: Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anupama Kizhakkeveettil, PhD, Principal Investigator — Southern California University of Health Sciences
Locations (1):
- Southern California University of Health Sciences, Whittier, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- SMTX: Any occurrence of SMT for cLBP in 2013, followed by initiation in 2013 of long-term management with OAT
- OATX: Any occurrence of OAT for cLBP in 2013, followed by initiation in 2013 of long-term management with SMT
Period: Overall Study
Arm/Group | Cohort SMT | Cohort OAT | SMTX | OATX
Started | 73 | 22 | 47 | 53
Completed | 73 | 22 | 47 | 53
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort SMT | Cohort OAT | Cohort SMTX | Cohort OATX | Total
Number analyzed (Participants) | 73 | 22 | 47 | 53 | 195
Age, Continuous [Mean (Standard Deviation); unit: years] | 78 (3.6) | 78 (3.7) | 78 (3.6) | 77 (4.1) | 78 (3.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Based on Medicare CMS data reporting guidelines, we are required by Data Use Agreement to suppress the data with small cell numbers ( DUA #).
  Here " 0"means data were not reported because cell numbers are suppressed by Medicare regulations
  Participants
    number analyzed (Participants) | 73 | 0 | 47 | 0 | 120
    Female | 54 | 0 | 33 | 0 | 87
    Male | 19 | 0 | 14 | 0 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Measure Analysis Population Description: Zero = not reported. Cell numbers are suppressed in accordance with Medicare regulations. Population: Based on Medicare CMS data reporting guidelines, we are required by Data Use Agreement to suppress the data with small cell numbers ( DUA #).
  Here Zero means data were not reported because cell numbers are suppressed by Medicare regulations.
  Participants
    number analyzed (Participants) | 71 | 19 | 45 | 50 | 185
    Hispanic or Latino | 0 | 0 | 0 | 0 | 0
    Not Hispanic or Latino | 71 | 19 | 45 | 50 | 185
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Self-reported QOL - Physical Health
Description: 1. Self-reported Quality of Life
  2. Scale range- There are 12 questions with scales of categorical values. Corresponding numeric values will be given to each category.
  3. Value range from "0" to "100"
  4. Higher scores reflecting better outcomes.
Time Frame: Base line. The survey (outcome measure) will be administered at at day one.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cohort SMT | Cohort OAT | Cohort SMTX | Cohort OATX
Number analyzed (Participants) | 73 | 22 | 47 | 53
units on a scale | 41.7 (11.2) | 28.8 (9.2) | 31.8 (8.7) | 32.9 (11.5)

2. Primary Outcome: Satisfaction With Care
Description: 1. Satisfaction with the Care
  2. The survey measured satisfaction for both SMT and PDT on a scale from 0-10, "0" being very dissatisfied and "10" being very satisfied. The patients were also given an option to select 'not applicable' if they never experienced either PDT or SMT.
  3. Higher numerical values indicate more satisfaction.
Time Frame: Base line.The survey (outcome measure) will be administered at day one.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Cohort SMT | Cohort OAT | Cohort SMTX | Cohort OATX
Number analyzed (Participants) | 73 | 22 | 47 | 53
Score on a scale | 8.9 (1.7) | 7.2 (2.5) | 4.9 (3.33) | 8.2 (2.5)

3. Primary Outcome: Beliefs Regarding Back Pain and Its Treatment
Description: 1. Beliefs about Treatments for Low Back Pain
  2. Scale range- Categorical values of Strongly disagree, Disagree, Undecided, Agree, Strongly agree (corresponding to numeric value 1, 2, 3, 4, and 5).
  3. For purposes of analysis, we combined the response options into the following three categories: "Disagree" (Strongly Disagree and Disagree), "Agree" (Strongly Agree and Agree), and "Undecided"(left as is).
  4. For interpreting the results for this scale, we reported only the number of people who agreed with the statements.
Time Frame: Base line.The survey (outcome measure) will be administered at at day one.
Population: Not every participant responded to all the questions. Results account for missing data.
Measure: Number; unit: participants number
Arm/Group | Cohort SMT | Cohort OAT | Cohort SMTX | Cohort OATX
Number analyzed (Participants) | 71 | 21 | 46 | 51
participants number
  Taking/having spinal manipulation for low back pain makes a lot of sense | 68 | 7 | 33 | 46
  Taking/having prescription drugs for low back pain makes a lot of sense | 9 | 19 | 23 | 16
  I think spinal manipulation is pretty useless for people with low back pain | 5 | 5 | 41 | 10
  I think taking prescription drugs are pretty useless for people with low back pain | 34 | 19 | 14 | 15
  I have concerns about taking/having spinal manipulation for my low back pain | 49 | 12 | 6 | 8
  I have concerns about taking/having prescription drugs for my low back pain | 53 | 5 | 23 | 29
  I am confident spinal manipulation would be suitable treatment for my low back pain | 64 | 5 | 31 | 41
  I am confident prescription drugs would be suitable treatment for my low back pain. | 7 | 19 | 23 | 12

ADVERSE EVENTS:
Time Frame: "Adverse Events were not monitored/assessed"
Description: "Adverse Events were not monitored/assessed"
Arm/Group | Cohort SMT | Cohort OAT | Cohort SMTX | Cohort OATX
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The overall response rate was lower than expected and we observed an age difference between respondents and non-respondents. In addition, recall bias is a potential limitation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-02): https://cdn.clinicaltrials.gov/large-docs/54/NCT03669354/Prot_SAP_000.pdf